CLINICAL TRIAL: NCT01377636
Title: Study to Measure BIS and Awareness in Patients Receiving Isoproterenol During Catheter Ablation for Atrial Fibrillation
Brief Title: Measurement of Bispectral Index and Awareness in Patients Undergoing Electrophysiology Studies With Isoproterenol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H#: 09-0440
Record Dates: First submitted 2010-03-22; First posted 2011-06-21 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Intraoperative Awareness
Keywords: Isoproterenol; Bispectral index (BIS); electrophysiology studies (EPS)
MeSH Terms: conditions — Intraoperative Awareness | interventions — Isoproterenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isoproterenol, BIS, forearm test (Experimental): 30 consecutive patients scheduled for EP studies under general anesthesia will participate in the study. Patients with neuromuscular disease precluding the use of succinylcholine will be excluded. The only other exclusions will be patient or cardiologist refusal. No attempts will be made to alter concurrent patient medication.
  Interventions: Drug: Isoproterenol

INTERVENTIONS:
Drug: Isoproterenol — patients will receive isoproterenol, have a BIS monitoring device and a modified isolated forearm test (no neuromuscular blockade).
  Other Names: isoprenaline

SUMMARY:
Isoproterenol is used as a cardiac stimulant in electrophysiology studies (EP). Preliminary data suggests that administration of isoproterenol increases the Bispectral index (BIS). BIS is used to monitor neuronal signals under anesthesia. The BIS level is suggested to correspond to the level of consciousness. We hypothesize that isoproterenol increases BIS values because it increases the patient's level of consciousness through its central nervous system (CNS) stimulatory effects. In this study, we will administer increasing doses of isoproterenol to EPS patients. We will measure the BIS levels continuously before and after isoproterenol administration. In addition, we will test the level of awareness of patients by their response to a modified isolated forearm technique.

DETAILED DESCRIPTION:
Isoproterenol is a direct acting Beta-1 and Beta-2 agonist useful for its effects on bronchodilation and myocardial contractility. Its CNS side effects include nervousness, headache, dizziness, restlessness, insomnia, anxiety, tension, blurring of vision, fear, and excitement. In addition to our preliminary data, two case reports show an increase in BIS with administration of isoproterenol. Our hypothesis is that administration of isoproterenol will increase the level of consciousness of the patient as reflected in the BIS reading.

The BIS Vista Monitor is a non-invasive device that measures the electrical activity of the brain. It computes a number between 0 and 100 which corresponds to a level of consciousness which is known as the Bispectral (BIS) value. Using the BIS value to guide administration of anesthetic medication, clinicians can make informed decisions for optimal anesthesia. This technology has the potential to prevent over sedation, but is currently not a standard monitoring device.

Another approach to evaluating the level of consciousness of anesthetized patients is to assess their ability to form memories or recall events which occurred while under anesthesia. Conscious recall is the first to disappear with decreasing levels of consciousness. A BIS of 60 or less has been shown in various studies to be sufficient to prevent conscious recall in the vast majority of patients. We propose to use a modified isolated forearm technique test in which the patient is asked to squeeze an observer's hand during anesthesia to ascertain if awareness can occur without recall at a BIS of 60 to 70. (6) Implicit memory in which there is no conscious recall or evaluation of awareness can be assessed by word stem completion tests and has been shown to occur with a BIS as low as 40 - 60 although these results are not consistent across all studies. (7)

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for EP studies for catheter ablation of atrial fibrillation under general anesthesia will participate in the study

Exclusion Criteria:

* Patients with neuromuscular disease precluding the use of succinylcholine will be excluded.
* Patient or cardiologist refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Linton, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, Department of Anesthesiology, New York, New York, United States

REFERENCES:
- [Background] O'Neill DK, Aizer A, Linton P, Bloom M, Rose E, Chinitz L. Isoproterenol infusion increases level of consciousness during catheter ablation of atrial fibrillation. J Interv Card Electrophysiol. 2012 Aug;34(2):137-42. doi: 10.1007/s10840-011-9652-3. Epub 2012 Feb 25. PMID 22366997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the preoperative evaluation for anesthesia, the patients scheduled for catheter ablation for atrial fibrillation were approached by the research associate for informed consent and enrollment into the study. The research consent was separate from the clinical anesthesia and procedural consents.
Groups:
- Pre and Post Isoproterenol Infusion: Bispectral EEG (BIS) monitoring and neurological examinations were repeated throughout an isoproterenol infusion protocol (20 minutes maximum) to measure the changes in arousal and ability to follow commands under anesthesia
Period: Overall Study
Arm/Group | Pre and Post Isoproterenol Infusion
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre and Post Isoproterenol Infusion: Subjects undergoing catheter ablation for atrial fibrillation had measurements pre and post isoproterenol infusion
Arm/Group | Pre and Post Isoproterenol Infusion
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants] — Demographics and BIS were measured
  Participants
    <=18 years | 0
    Between 18 and 65 years | 11
    >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Increase in BIS Readings During Steady State
Description: Increasing doses of isoproterenol (5,10,15,20 mcg/minute) were administered to patients undergoing catheter ablation for atrial fibrillation. BIS levels were measured continuously before and after isoproterenol administration. Number of participants with increase in BIS reading during anesthetic steady state are reported below. The BIS scale ranges from 0 to 100. The individual's baseline BIS was measured continuously and was maintained in an anesthetic steady state with minimum variance prior to isoproterenol. A deviation from the mean in excess of 3 points (2 STD) was defined categorically as a positive response and was counted dichotomously.
Time Frame: During time of Electrophysiology (EP) studies.
Measure: Number; unit: participants
Groups:
- Pre and Post Isoproterenol Infusion: BIS monitoring and neurological examinations were repeated throughout an isoproterenol infusion protocol (20 minutes maximum) to measure the changes in arousal and ability to follow commands under anesthesia
Arm/Group | Pre and Post Isoproterenol Infusion
Number analyzed (Participants) | 20
participants | 19

2. Secondary Outcome: Number of Participants With Spontaneous Musculoskeletal Movement
Description: Increasing doses of isoproterenol (5,10,15,20 mcg/minute) were administered to patients undergoing catheter ablation for atrial fibrillation. Patients under steady state total venous anesthesia (TIVA) with propofol and remifentanil infusions with BIS around 50 normally do not move even in the absence of neuromuscular blockade. Spontaneous movement appearing like restlessness during sleep is unusual. Several patients under anesthesia after isoproterenol appear to wake up and move spontaneously.
Time Frame: Within 20 minutes of starting isoproterenol infusion
Measure: Number; unit: participants
Arm/Group | Isoproterenol, BIS, Forearm Test
Number analyzed (Participants) | 20
participants | 12

3. Secondary Outcome: Number of Participants Who Follow Verbal Command to Squeeze Hands
Description: Increasing doses of isoproterenol (5,10,15,20 mcg/minute) were administered to patients undergoing catheter ablation for atrial fibrillation. Ability to follow verbal commands before and after isoproterenol infusion was assessed by asking subjects to "squeeze my hands".
Time Frame: Within 20 minutes of starting isoproterenol infusion
Measure: Number; unit: participants
Arm/Group | Isoproterenol, BIS, Forearm Test
Number analyzed (Participants) | 20
participants | 10

4. Other Pre Specified Outcome: Number of Participants With Significant Change in Heart Rate
Description: Heart rate measured by standard EKG monitor during anesthesia. Pre- and Post Heart rates where noted. An increase of 8 percent or more was defined as a significant change in heart rate.
Time Frame: Within 20 minutes of starting isoproterenol infusion
Measure: Number; unit: participants
Arm/Group | Pre and Post Isoproterenol Infusion
Number analyzed (Participants) | 20
participants | 18

5. Other Pre Specified Outcome: Number of Participants With Change in Blood Pressure
Description: Non-Invasive Blood Pressure (NIBP) is measured routinely as part of an anesthetic. Pre- and Post Blood Pressures where noted. An increase or decrease of 10 percent or more was defined as a significant change in systolic blood pressure.
Time Frame: Within 20 minutes of starting isoproterenol infusion
Measure: Number; unit: participants
Arm/Group | Pre and Post Isoproterenol Infusion
Number analyzed (Participants) | 20
participants | 13

6. Other Pre Specified Outcome: Number of Participants With Amnesia or No Recall During Steady State
Description: Increasing doses of isoproterenol (5,10,15,20 mcg/minute) were administered to patients undergoing catheter ablation for atrial fibrillation. Specific pre-determined test words were spoken to the subject during administration of isoproterenol. After anesthesia, patients were tested for possible recall of those specific words. If no words were recalled, the result was categorically defined as amnesia.
Time Frame: Within one hour of completing anesthesia
Measure: Number; unit: participants
Arm/Group | Isoproterenol, BIS, Forearm Test
Number analyzed (Participants) | 20
participants | 20

7. Other Pre Specified Outcome: Number of Participants With New Arrhythmia During Steady State.
Description: Increasing doses of isoproterenol (5,10,15,20 mcg/minute) were administered to patients undergoing catheter ablation for atrial fibrillation after return to sinus rhythm. If a non-sinus arrhythmia resulted from the infusion, the arrhythmia was defined categorically as a positive response and was counted dichotomously.
Time Frame: Within 20 minutes of start of isoproterenol
Measure: Number; unit: participants
Arm/Group | Pre and Post Isoproterenol Infusion
Number analyzed (Participants) | 20
participants | 4

8. Other Pre Specified Outcome: Number of Participants Who Developed Ischemia or ST Segment Changes
Description: The (ST) segment on the EKG was monitored for changes suggestive of demand ischemia. An observable EKG change compared to baseline was defined categorically as a positive response and was counted dichotomously.
Time Frame: Within 20 minutes of starting isoproterenol infusion
Measure: Number; unit: participants
Arm/Group | Pre and Post Isoproterenol Infusion
Number analyzed (Participants) | 20
participants | 2

9. Primary Outcome: BIS Change
Description: The BIS scale ranges from 0 to 100. The individual's baseline BIS was measured continuously and was maintained in an anesthetic steady state with minimum variance prior to isoproterenol. A deviation from the mean in excess of 3 points (2 STD) was defined categorically as a positive response and was counted dichotomously.The difference between Pre-BIS and Post-BIS was calculated.
Time Frame: Within 20 minutes of starting isoproterenol infusion
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pre and Post Isoproterenol Infusion
Number analyzed (Participants) | 20
units on a scale | 24.6 [19.3 to 29.9]

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Pre and Post Isoproterenol Infusion: In this study, serious adverse events were considered clinically significant adverse events. The well known isoproterenol effects on heart rate, rhythm, ST segments, and blood pressure were noted.
Arm/Group | Pre and Post Isoproterenol Infusion
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre and Post Isoproterenol Infusion (N=20)
Death (Cardiac disorders) | 0 (0)
Stroke (Nervous system disorders) | 0 (0)
Seizure (Nervous system disorders) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre and Post Isoproterenol Infusion (N=20)
Tachycardia (Cardiac disorders) | 19 (19) — Elevated heart rate
Atrial Fibrillation/Junctional Rhythm (Cardiac disorders) | 4 (4) — Non-Sinus Rhythm
ST Changes (transient) (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 6 (6) — Decrease in Systolic Blood Pressure more than 20 mm Hg
Hypertension (Cardiac disorders) | 6 (6) — Increase of Systolic Blood Pressure in excess of 20 mm Hg
Bradycardia (Cardiac disorders) | 0 (0) — Decrease in Heart Rate below 60
Ventricular arrhythmia (Cardiac disorders) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0)
Bleeding (Blood and lymphatic system disorders) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No